CLINICAL TRIAL: NCT06558968
Title: Evaluation of Polyetheretherketone and Monolithic Zirconia as Esthetic Functional Space Maintainers in Children (A Randomized Clinical Trial)
Brief Title: Evaluation of PEEK and BruxZir as Esthetic Space Maintainers in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hagar Abozeid, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PED21-8D
Record Dates: First submitted 2021-08-30; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Dentistry

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: articipants will be blinded to the type of intervention. Teeth treated will be assigned codes so that outcome evaluators at the follow up appointments are blinded. On the other hand, the operator/ primary investigator cannot be blinded, as she is already familiar with the nature of the materials used. For statistical analysis, codes will also assure blinding and confidentiality. For the patient, both types of space maintainers will have the same color and design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polyetheretherketone (Active Comparator): PEEK 'Polyetheretherketone' Victrex® is a type of polymer with suitable mechanical and
  physical properties. It is a resilient material with high flexural strength and resistance
  to deformation. Therefore, it can be used in fixed prosthesis and space maintainers
  Interventions: Other: aesthetic functional space maintainers
- monolithic zirconia (Active Comparator): BruxZir® is a type of monolithic zirconia with higher flexural strength and fracture toughness than the classic zirconia and can withstand the changes in temperature in the oral cavity. Therefore it can be used as a space maintainer
  Interventions: Other: aesthetic functional space maintainers

INTERVENTIONS:
Other: aesthetic functional space maintainers — evaluate the use of Polyetheretherketone 'PEEK' and monolithic zirconia 'Bruxzir' as esthetic functional band and loop space maintainers.

SUMMARY:
Compare two band and loop space maintainers made from two tooth colored materials; Polyetherethherketone (PEEK) and monolithic Zirconia (BruxZir) as regards to:

* Clinical performance of space maintainers in terms of frequency of debonding or fracture of the appliance and health of adjacent gingiva during a one-year follow up.
* Wear of the opposing teeth.

DETAILED DESCRIPTION:
After extraction of the mandibular first primary molars in both mandibular quadrants, impressions will be taken with intraoral scanner. Then, it will be sent to the CAD/CAM laboratory to construct functional band and loop space maintainers using PEEK and monolithic zirconia 'BruxZir' blocks with proper shades.

After the fabrication of the space maintainers of both sides, they will be cemented with resin luting cement containing MDP monomer. Photographs will be taken after cementation for the space maintainers and the patient will be informed and educated about the oral hygiene measures. The parents will also be inquired to call if any discomfort, debonding or fracture of the appliances happens.

ELIGIBILITY:
Inclusion Criteria:

* Clinical inclusion criteria:

  * Children requiring bilateral extraction of mandibular first primary molars or those with previously extracted molars no more than 6 months prior to intervention (11) .
  * Existence of teeth on the mesial and distal side of edentulous area.
  * Angle's Class I molar relationship and/or flush terminal/mesial step primary molar occlusion

Radiographic inclusion criteria:

* No periapical and/ or furcural pathological condition related to abutment teeth.
* Presence of tooth germ of the succeeding tooth (mandibular first premolars).
* Presence of more than 1 mm of bone overlying the successor tooth germ

Exclusion Criteria:

* Carious abutment teeth requiring pulp therapy.

  * Carious abutment primary teeth requiring a full coverage restoration.
  * Patients with history of bruxism or/and clenching.
  * Patients with medical, intellectual or physical disabilities.
  * Patients with abnormalities as posterior cross-bite, open bite, and deep bite

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Clinical performance | 1 year
  regarding debonding or fracture of the appliance. if debonding or fracture occur then this means failure.
Gingival health | 1 year
  Gingival Index of Loe and Silness. where score 0 indicates normal gingiva, score 1 mild inflammation (slight change in color, slight edema but no bleeding on probing. score 2 indicates moderate inflammation (redness, edema, bleeding on probing and score 3 refers to severe inflammation (marked redness, edema, ulceration with sponatnoeus bleeding.

SECONDARY OUTCOMES:
Wear of the opposing tooth | 1 year
  using CAD/CAM software Cerec software (Cerec 4.2, DentsplySirona, Bensheim, Germany)volumetric loss on the surfaces were calculated in the last follow up visit after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Khattab, Professor, Study Director — Ainshams U
Locations (1):
- Ain Shams University, Cairo, Egypt